CLINICAL TRIAL: NCT07123259
Title: Anti-Ulcerative Colitis Activity of Pomegranate (Punica Granatum L.) Peel Powder Muffins in Patients With Gastric Ulcer
Brief Title: Ulcer Pomegranate Muffins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sana Noreen, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC-UOL-/530/08/24
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-08

CONDITIONS: Gastric; Peptic Ulcer
Keywords: Punica granatum; Gastric Ulcer; Ulcerative Colitis; Helicobacter pylori
MeSH Terms: conditions — Peptic Ulcer; Stomach Ulcer; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment 1 group: Whole wheat muffin enriched with pomegranate peel powder (PPP=1.5g) (Active Comparator)
  Interventions: Combination Product: 1.5g enriched pomegranate muffins
- Treatment 2 group: Whole wheat muffin enriched with pomegranate peel powder (PPP=3g) (Active Comparator)
  Interventions: Combination Product: 3g enriched pomegranate muffins
- Group T0: Whole wheat muffin (Placebo Comparator): 400g whole wheat flour was used to formulate the muffins
  Interventions: Dietary Supplement: WHOLE WHEAT MUFFIN

INTERVENTIONS:
Dietary Supplement: WHOLE WHEAT MUFFIN — 400g whole wheat flour was used for the development of muffins
  Arms: Group T0: Whole wheat muffin
Combination Product: 1.5g enriched pomegranate muffins — 1.5 g of pomegranate peel powder (PPP), alongside conventional medical therapy
  Arms: Treatment 1 group: Whole wheat muffin enriched with pomegranate peel powder (PPP=1.5g)
Combination Product: 3g enriched pomegranate muffins — 3 g of pomegranate peel powder (PPP), alongside conventional medical therapy
  Arms: Treatment 2 group: Whole wheat muffin enriched with pomegranate peel powder (PPP=3g)

SUMMARY:
Pomegranate (Punica granatum L.) peel powder, known for its potent antioxidant, anti-inflammatory, and antimicrobial properties, has shown promise in the dietary management of gastrointestinal disorders. In recent clinical observations, incorporating pomegranate peel powder into muffins consumed by patients with gastric ulcers demonstrated potential anti-ulcerative colitis activity. The bioactive compounds in the peel, such as polyphenols (punicalagins, ellagic acid), help reduce oxidative stress and modulate inflammatory pathways in the gut. Patients consuming these enriched muffins reported improvements in gastrointestinal symptoms, reduced mucosal inflammation, and enhanced mucosal healing, suggesting a supportive role of pomegranate peel as a functional food ingredient in managing gastric and colitis-related conditions.

DETAILED DESCRIPTION:
2. Materials and Methods 2.1. Ethical Statement The study received ethical approval from the Research Ethics Committee (REC) of the University of Lahore (REC-UOL-/530/08/24). Informed consent was obtained from all participants, who were fully informed about the study's aims, methods, risks, and benefits, and were given the opportunity to ask questions and withdraw at any time.

2.2. Settings The research was undertaken at Umair Clinic, Gondal Chowk, Kacha Jail Road, Lahore, whereas laboratory work and muffin preparation were done at the Food Science and Nutrition Laboratory (FASH Lab 502), UIDNS, The University of Lahore, Lahore, Pakistan.

2.3. Subjects A randomized controlled trial (RCT) was conducted using a purposive sampling strategy. Initially, 88 patients were enrolled, accounting for a projected 20% dropout rate. One patient was excluded for not meeting the inclusion criteria, resulting in 87 eligible participants. These were randomly and equally assigned into three groups, with 29 patients in each group. During the study, two patients were excluded from the placebo Group (T0), leaving 27 participants. In Group 2 (T1), two patients were excluded, and one participant voluntarily withdrew due to personal health issues from Group 3 (T2). Ultimately, a total of 82 patients completed the 8-week trial study.

2.4. Intervention groups Group T1 received one muffin per day enriched with 1.5 g of pomegranate peel powder (PPP), alongside conventional medical therapy. Group T2 received two PPP-enriched muffins per day (totaling 3 g of PPP), in addition to conventional therapy. The placebo group received one whole wheat muffin per day without PPP supplementation. All participants consumed their assigned muffins once daily for 8 weeks 2.4.1 Demographic Profile Demographic data among ulcer patients, including age, gender, and socioeconomic status, were collected at baseline using a structured questionnaire (Saber et al., 2021).

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients aged 45-60 years with confirmed Helicobacter pylori
* infection verified through a stool antigen test (pH 7.0-7.5)
* elevated levels of pepsinogen I and II

Exclusion Criteria:

* pregnancy or lactation
* history of gastric surgery
* current use of proton pump inhibitors (PPIs)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Pepsinogen I and II Levels | 8 WEEKS
  Pepsinogen I and II levels were measured using an enzyme-linked immunosorbent assay (ELISA). These biomarkers were assessed to evaluate gastric mucosal integrity, with elevated levels indicating gastric inflammation and aiding in the diagnosis and monitoring of ulcer severity and progression (Zhang et al., 2024).
Helicobacter pylori Test | 8 WEEKS
  Pepsinogen I and II levels were measured using an enzyme-linked immunosorbent assay (ELISA). These biomarkers were assessed to evaluate gastric mucosal integrity, with elevated levels indicating gastric inflammation and aiding in the diagnosis and monitoring of ulcer severity and progression (Zhang et al., 2024).

SECONDARY OUTCOMES:
Complete blood count | 8 Weeks
  A complete blood count (CBC) was conducted using an automated hematology analyzer on EDTA-anticoagulated blood samples. Key parameters such as hemoglobin, RBC, WBC and platelet count were evaluated (Saleska et al., 2024).
Liver function assay | 8 Weeks
  Serum AST, ALT, and ALP were measured using an enzymatic colorimetric technique (Jalili et al., 2022).
Barium Test | 8 Weeks
  A barium swallow test was performed using oral barium sulfate and X-ray imaging to detect ulcers and structural abnormalities in the upper gastrointestinal tract (Kusano et al., 2024)

CONTACTS AND LOCATIONS:
Locations (1):
- Sana Noreen, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the Individual Participant Data (IPD) collected during the study with other qualified researchers upon reasonable request. The shared data will include de-identified participant-level data related to baseline characteristics, intervention, outcomes, and adverse events.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Kamali M, Tavakoli H, Khodadoost M, Daghaghzadeh H, Kamalinejad M, Gachkar L, Mansourian M, Adibi P. Efficacy of the Punica granatum peels aqueous extract for symptom management in ulcerative colitis patients. A randomized, placebo-controlled, clinical trial. Complement Ther Clin Pract. 2015 Aug;21(3):141-6. doi: 10.1016/j.ctcp.2015.03.001. Epub 2015 Apr 1. PMID 26256131